CLINICAL TRIAL: NCT04762628
Title: Randomized Trial to Assess the Efficacy and Safety of Dietary Supplements MAF Capsules, 148 mg and M Capsules, 148 mg in Addition to the Standard of Care (SOC) Compared SOC in the Treatment of Hospitalized With COVID-19 Patients Who Not Requiring the Mechanical Ventilation
Brief Title: Trial Efficacy of Saisei Pharma Dietary Supplements MAF Capsules, 148 mg and M Capsules, 148 mg in Hospitalized COVID-19 Patients
Acronym: SaiseiCovUKR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saisei Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SaiseiMAF supplements COVID
Record Dates: First submitted 2021-02-11; First posted 2021-02-21 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Covid19
Keywords: Covid19; Colostrum MAF; Supplements; Oxygen supply; Mortality; Clinical improvement; lymphocyte depletion prevention
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MAF capsules (Experimental): MAF capsules 148 mg TID for 14 days + Standard of care
  Interventions: Dietary Supplement: MAF capsules 148 mg
- M capsules (Experimental): M capsules 148 mg TID for 14 days + Standard of care
  Interventions: Dietary Supplement: M capsules 148 mg
- Comparison (Active Comparator): Standard of care
  Interventions: Other: Standard of care

INTERVENTIONS:
Dietary Supplement: MAF capsules 148 mg — enteric capsules based on enzymatically treated bovine colostrum
  Arms: MAF capsules
Dietary Supplement: M capsules 148 mg — enteric capsules based on enzymatically treated bovine whey
  Arms: M capsules
Other: Standard of care — Standard of care
  Arms: Comparison

SUMMARY:
The SaiseiCovUKR clinical study is a multicentric, randomized trial study targeting patients hospitalized with COVID-19 who do not require mechanical ventilation. This study aims to provide preliminary data on the activity and safety of MAF capsules and M capsules in the target population after 14 days of dosing. MAF capsules and M capsules are dietary supplements targeting the gut's mucosal immunity to control local and systemic inflammation, limiting epithelial damage and preventing the accumulation of pathological macrophage populations at sites of SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Saisei Pharma is developing biologics using an enzymatic modification of Vitamin D binding protein and other glycoproteins in biological substrates, which have been shown to increase macrophage phagocytic and antigen processing activity without promoting the proinflammatory profile of macrophages. Bovine colostrum is the substrate for MAF capsules and bovine whey for M capsules. The enteric capsules formulation of the investigational dietary supplements is targeting the gut mucosa and its associated natural anti-inflammatory macrophages profile. The SaiseiCovUKR clinical study is multicentric, randomized, open-label in hospitalized patients with moderate and severe COVID-19 to provide data on the activity and safety of MAF capsules and M capsules in the target population after 14 days of dosing. The trial will use an adaptive design based on a pre-specified criteria, using an independent external Data Monitoring Committee (DMC) to monitor safety, efficacy, and review data at appropriate intervals. The general objectives of the study are to obtain a preliminary indication of activity of MAF capsules and M capsules on shortened time to recovery and decreased mortality in the target population (600 patients, age ≥ 18 years). The study results can provide a background for further investigation of the studied dietary supplements as new drugs in COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Patients found to have positive RT-PCR for SARS-CoV-2 in any specimen on 4 days prior to randomization, those who are hospitalized with evidence of respiratory disease during clinical assessment or imaging
2. Male or non-pregnant female adult ≥18 years of age subject (or legally authorized representative) provides informed consent prior to initiation of any study procedures
3. Subject (or legally authorized representative) understands and agrees to comply with planned study procedures
4. Has illness of not more than 7 days duration
5. At the time of enrolment does not require immediate resuscitation or mechanical ventilation
6. Respiration rate ≤ 29 per minute
7. SpO2 ≤ 95% on room air
8. Agrees to not participate in another clinical trial through Day 29

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Known allergy to dairy products
3. On corticosteroids for COVID-19 therapy at the time of screening
4. Subjects who are taking corticosteroids or other immunosuppressive drugs for other medical conditions
5. Concurrent malignancy requiring chemotherapy
6. Known renal insufficiency with glomerular filtration rate (eGFR) < 30 ml/min (including patients receiving hemodialysis or hemofiltration).
7. ALT or AST > 5 times the upper limit of normal
8. Subjects receiving other immune-based therapy for COVID-19, such as convalescent plasma, immunoglobulin products, interferons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
The time to basic clinical improvement and to recovery defined as the following | Day 1 through Day 29
  * Hospitalized, not requiring supplemental oxygen, requires ongoing medical care
  * Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care
  * Not hospitalized, limitation on activities and/or requiring home oxygen
  * Not hospitalized, no limitations on activities
14-day Participant Mortality | Day 1 through Day 14
  The mortality rate will be determined as the proportion of participants who died by study Day 14
29-day Participant Mortality | Day 1 through Day 29
  The mortality rate will be determined as the proportion of participants who died by study Day 29

SECONDARY OUTCOMES:
Percentage of Participants in Each Clinical Status Category as Assessed by a 9-Point Ordinal Scale on Day 14 | Day 14
  Clinical status derives from death, hospital discharge, and 9-Point Ordinal Scale as follows: score of "8" use for all days on or after the date of death; score of "0" use for all days on or after discharged alive date; last available assessment for missing value. The scale is as follows: 8. Death; 7. Hospitalized, on invasive mechanical ventilation with vasopressor or Extracorporeal Membrane Oxygenation; 6. Hospitalized, on invasive mechanical ventilation; 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring low flow supplemental oxygen; 3. Hospitalized, not requiring supplemental oxygen - requires ongoing medical care (coronavirus (COVID-19) related or otherwise; 2. Not hospitalized, limitation on activities and/or requiring home oxygen; 1. Not hospitalized, no limitation on activities; 0. No clinical or virological evidence of infection
Time to an improvement of one category from admission on 9-Point Ordinal Scale | Day 1 through Day 29
  Time to reach an improvement of one category from admission on 9-Point Ordinal Scale. The scale is as follows: 8. Death; 7. Hospitalized, on invasive mechanical ventilation with vasopressor or Extracorporeal Membrane Oxygenation; 6. Hospitalized, on invasive mechanical ventilation; 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring low flow supplemental oxygen; 3. Hospitalized, not requiring supplemental oxygen - requires ongoing medical care (coronavirus (COVID-19) related or otherwise; 2. Not hospitalized, limitation on activities and/or requiring home oxygen; 1. Not hospitalized, no limitation on activities; 0. No clinical or virological evidence of infection
Time to an improvement of two categories from admission on 9-Point Ordinal Scale | Day 1 through Day 29
  Time to reach an improvement of two categories from admission on 9-Point Ordinal Scale. The scale is as follows: 8. Death; 7. Hospitalized, on invasive mechanical ventilation with vasopressor or Extracorporeal Membrane Oxygenation; 6. Hospitalized, on invasive mechanical ventilation; 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring low flow supplemental oxygen; 3. Hospitalized, not requiring supplemental oxygen - requires ongoing medical care (coronavirus (COVID-19) related or otherwise; 2. Not hospitalized, limitation on activities and/or requiring home oxygen; 1. Not hospitalized, no limitation on activities; 0. No clinical or virological evidence of infection
Percentage of Participants in Each Clinical Status Category as Assessed by a 9-Point Ordinal Scale on Day at days 3, 5, 8, 11,14 and 29 | Days 3, 5, 8, 11,14 and 29
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8. Death; 7. Hospitalized, on invasive mechanical ventilation with vasopressor or Extracorporeal Membrane Oxygenation; 6. Hospitalized, on invasive mechanical ventilation; 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring low flow supplemental oxygen; 3. Hospitalized, not requiring supplemental oxygen - requires ongoing medical care (coronavirus (COVID-19) related or otherwise; 2. Not hospitalized, limitation on activities and/or requiring home oxygen; 1. Not hospitalized, no limitation on activities; 0. No clinical or virological evidence of infection
Mean change in the ranking on 9-Point Ordinal Scale from baseline to days 3, 5, 8, 11, 14 and 29 | Days 3, 5, 8, 11, 14 and 29
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8. Death; 7. Hospitalized, on invasive mechanical ventilation with vasopressor or Extracorporeal Membrane Oxygenation; 6. Hospitalized, on invasive mechanical ventilation; 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring low flow supplemental oxygen; 3. Hospitalized, not requiring supplemental oxygen - requires ongoing medical care (coronavirus (COVID-19) related or otherwise; 2. Not hospitalized, limitation on activities and/or requiring home oxygen; 1. Not hospitalized, no limitation on activities; 0. No clinical or virological evidence of infection
Duration of conventional oxygen therapy Use | Day 1 through Day 29
  Duration of conventional oxygen therapy use measured in days among participants who were on conventional oxygen therapy use at baseline
Duration of new conventional oxygen therapy use | Day 1 through Day 29
  Duration of new conventional oxygen therapy use measured in days among participants who were not on conventional oxygen therapy use at baseline
Duration of Non-invasive Ventilation or High Flow Oxygen Use | Day 1 through Day 29
  Duration of non-invasive ventilation or high flow oxygen use measured in days among participants who were on non-invasive ventilation or high-flow oxygen use at baseline
Duration of New Non-invasive Ventilation or High Flow Oxygen Use | Day 1 through Day 29
  Duration of new non-invasive ventilation or high flow oxygen use measured in days among participants who were not on non-invasive ventilation or high-flow oxygen use at baseline
Duration of Mechanical Ventilator or Extracorporeal Membrane Oxygenation (ECMO) Use | Day 1 through Day 29
  Duration of Mechanical Ventilator or ECMO Use in days among all participants to whom it will be administrated
Percentage of Participants Requiring New Oxygen Use | Day 1 through Day 29
  The percentage of participants requiring new oxygen determined as the percentage of participants not requiring oxygen at baseline
Percentage of Participants Requiring New Non-invasive Ventilation or High-flow Oxygen Use | Day 1 through Day 29
  New non-invasive ventilation or high-flow oxygen use determined as the percentage of subjects not on non-invasive ventilation or high-flow oxygen at baseline.
Percentage of Participants Requiring Ventilator or ECMO Use | Day 1 through Day 29
  The percentage of participants requiring Ventilator or ECMO Use
Incidents of post-COVID-19 related symptoms at Day 29 | Day 29
  Incidents of all post-COVID-19 symptoms, which will be reported in the post-COVID-19 questionnaire form
Incidents of post-COVID-19 related symptoms at Day 60 | Day 60
  Incidents of all post-COVID-19 symptoms, which will be reported in the post-COVID-19 questionnaire form
Percentage of participants with post-COVID-19 related symptoms at Day 29 | Day 29
  Percentage of participants with presents post-COVID-19 related symptoms
Percentage of participants with post-COVID-19 related symptoms at Day 60 | Day 60
  Percentage of participants with presents post-COVID-19 related symptoms
Percentage of Participants Reporting Grade 3 and 4 Clinical and/or Laboratory Adverse Events (AEs) | Day 1 through Day 29
  Grade 3 AEs are defined as events interrupting daily living activities, or significantly affecting clinical status, or requiring intensive therapeutic intervention. Severe events are usually incapacitating. Grade 4 AEs are defined as potentially life threatening.
Percentage of Participants Reporting Serious Adverse Events (SAEs) | Day 1 through Day 29
  An SAE is defined as an AE or a suspected adverse reaction is considered serious if, in the view of either the investigator or the sponsor, it results in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
Percentage of Participants Discontinued or Temporarily Suspended From Investigational dietary supplements | Day 1 through Day 14
  Participants may have discontinued from investigational dietary supplements due to product intolerability, applied mechanical ventilation, swallowing impairment, or death. The discontinuation or temporary suspension intake of studied supplements for any reason will be collected.
Change From Baseline in Alanine Transaminase (ALT) | Days 1, 7, 14 and 29
  To evaluate ALT, blood will be collected at Days 1, 7, and 14 while participants are inpatient, and at Day 29, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge.
Change From Baseline in Aspartate Transaminase (AST) | Days 1, 7, 14 and 29
  To evaluate AST, blood will be collected at Days 1, 7, and 14 while participants are inpatient, and at Day 29, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge.
Change From Baseline in Total Bilirubin | Days 1, 7, 14 and 29
  To evaluate Total Bilirubin, blood will be collected at Days 1, 7, and 14 while participants are inpatient, and at Day 29, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge.
Change From Baseline in Creatinine | Days 1, 7, 14 and 29
  To evaluate serum Creatinine, blood will be collected at Days 1, 7, and 14 while participants are inpatient, and at Day 29, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge.
Change From Baseline in Glucose | Days 1, 7, 14 and 29
  To evaluate serum Glucose, blood will be collected at Days 1, 7, and 14 while participants are inpatient, and at Day 29, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge.
Change From Baseline in Hemoglobin | Days 1, 7, 14 and 29
  To evaluate Hemoglobin, blood will be collected at Days 1, 7, and 14 while participants are inpatient, and at Day 29, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge.
Change From Baseline in Platelets | Days 1, 7, 14 and 29
  To evaluate Platelets, blood will be collected at Days 1, 7, and 14 while participants are inpatient, and at Day 29, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge.
Change From Baseline in White Blood Cell Count (WBC) | Days 1, 7, 14 and 29
  To evaluate WBC, blood will be collected at Days 1, 7, and 14 while participants are inpatient, and at Day 29, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge.
Change From Baseline in Lymphocytes | Days 1, 7, 14 and 29
  To evaluate Lymphocytes, blood will be collected at Days 1, 7, and 14 while participants are inpatient, and at Day 29, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge.

OTHER OUTCOMES:
Change From Baseline in C-Reactive Protein | Days 1, 7 and 14
  To evaluate C-Reactive Protein, blood will be collected at Days 1, 7 and 14 while participants are inpatient, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge
Change From Baseline in D-Dimer | Days 1, 7 and 14
  To evaluate D-Dimer, blood will be collected at Days 1, 7 and 14 while participants are inpatient, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge
Change From Baseline in Lactate Dehydrogenase | Days 1, 7 and 14
  To evaluate Lactate Dehydrogenase, blood will be collected at Days 1, 7 and 14 while participants are inpatient, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge
Change From Baseline in Ferritin | Days 1, 7 and 14
  To evaluate Ferritin, blood will be collected at Days 1, 7 and 14 while participants are inpatient, with the Day 1 assessment serving as the baseline. Participants who will be discharged will have blood collected if infection control measures allow in-person visits after discharge

CONTACTS AND LOCATIONS:
Locations (2):
- Ukraine (2):
  - The Central Hospital of Rubizhne, Infection Disease Department, Rubizhne, Luhansk Oblast
  - Municipal Kharkiv Regional Infectious Diseases Clinical Hospital, Kharkiv

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared via ISARIC COVID-19 Clinical Database.
Time Frame: Request for data will be indefinitely available
Access Criteria: Reasonable request to investigators

REFERENCES:
- [Background] Kawakatsu K, Ishikawa M, Mashiba R, Tran NK, Akamatsu M, Nishikata T. Characteristic Morphological Changes and Rapid Actin Accumulation in Serum-MAF-treated Macrophages. Anticancer Res. 2019 Aug;39(8):4533-4537. doi: 10.21873/anticanres.13630. PMID 31366556
- [Background] Uto Y, Kawai T, Sasaki T, Hamada K, Yamada H, Kuchiike D, Kubo K, Inui T, Mette M, Tokunaga K, Hayakawa A, Go A, Oosaki T. Degalactosylated/Desialylated Bovine Colostrum Induces Macrophage Phagocytic Activity Independently of Inflammatory Cytokine Production. Anticancer Res. 2015 Aug;35(8):4487-92. PMID 26168491
- [Background] Greilberger J, Herwig R. Vitamin D - Deglycosylated Vitamin D Binding Protein Dimer: Positive Synergistic Effects on Recognition, Activation, Phagocytosis and Oxidative Stress on Macrophages. Clin Lab. 2020 Jan 1;66(1). doi: 10.7754/Clin.Lab.2019.191121. PMID 32013346
- [Derived] Inui T, Kruglova O, Martynenko O, Martynenko K, Tieroshyn V, Gavrylov A, Kubo K, Yamakage H, Kutsyn B, Kubashko A, Veklych Z, Terashima Y, Mette M, Kutsyna G. Effect of degalactosylated bovine glycoprotein formulations MAF and M small es, Cyrillicapsules on lymphopenia and clinical outcomes in hospitalized COVID-19 patients: a randomized clinical trial. BMC Infect Dis. 2024 May 23;24(1):519. doi: 10.1186/s12879-024-09286-0. PMID 38783176